CLINICAL TRIAL: NCT03043352
Title: Evaluation of the Effectiveness and Impact of Community Case Management of Severe Acute Malnutrition Through Lady Health Workers As Compared To a Facility Based Program: A Cluster Randomized Controlled Trial
Brief Title: Evaluation of the Effectiveness and Impact of Community Case Management of Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Action Contre la Faim (Other)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3276-Ped-ERC-14
Record Dates: First submitted 2015-11-11; First posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Severe Malnutrition
Keywords: SAM; Malnutrition; LHW; CMAM
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (intervention) (Experimental): 'Management of SAM at home' LHWs will identify and treat all cases of severe acute malnutrition (SAM) as per the study eligibility criteria (MUAC < 11.5 cm) and manage all cases of SAM without complications at home with 'Standard CMAM program'. The LHWs will also identify SAM with complications for further assessment to the BHU Doctor and subsequent referral to the stabilization center . They will also provide one to one health and Infant and Young Child Feeding (IYCF) counselling to care takers of children in their catchment area.
  Interventions: Dietary Supplement: Management of SAM at home
- Group B (Control) (Active Comparator): 'Management of SAM at facility' LHWs will identify SAM as per 'Standard CMAM program' (MUAC < 11.5cm) and will refer all cases to the health facility BHU/ satellite site (ACF) for further management and counselling by health workers (ACF CMAM Nurse) at facility level.
  Interventions: Dietary Supplement: Management of SAM at facility

INTERVENTIONS:
Dietary Supplement: Management of SAM at home — LHWs will identify and treat all cases of severe acute malnutrition (SAM) in children under-five years at household level compared with the standard CMAM program
  Arms: Group A (intervention)
Dietary Supplement: Management of SAM at facility — LHWs will identify SAM as per 'Standard CMAM program' (MUAC < 11.5cm) and will refer all cases to the health facility BHU/ satellite site (ACF) for further management and counselling by health workers (ACF CMAM Nurse) at facility level.
  Arms: Group B (Control)

SUMMARY:
HYPOTHESIS:

Investigators hypothesize that by provision of care at household level in a community through lady health workers will as effective (recovery rate, burden of SAM, cost effective, coverage) as through health care providers at facility level. OBJECTIVES

1. To evaluate the effectiveness (rate of recovery, burden & coverage), of SAM standard management of children 06-59 months delivered at household level by first level health care providers (Lady health workers) compared with the standard CMAM program delivered at health facility by Govt./ACF staff.
2. To evaluate the cost effectiveness of treatment of SAM provided by LHWs at community level versus treatment delivered at health facility by Govt/ACF staff.

STUDY DESIGN:

Cluster randomized controlled trial

SAMPLE SIZE & RANDOMIZATION:

Investigators took 6% prevalence to calculate the sample size with an expected reduction of 20%. A sample size of 3 clusters per group with 150 individuals per cluster is needed. STUDY METHODOLOGY Intervention (Group A): LHWs will identify and treat all cases of severe acute malnutrition (SAM) as per the study eligibility criteria (MUAC < 11.5 cm) and manage all cases of SAM without complications at home following the national CMAM guidelines. Control (Group B): LHWs will identify SAM as per the CMAM guidelines (MUAC < 11.5 cm) and will refer all cases to the health facility (ACF) for further management and counselling by health workers at facility.

DETAILED DESCRIPTION:
INTRODUCTION & RATIONALE:

There is good evidence of the success of CMAM programs for treating SAM in emergencies and humanitarian crises [1], but little regarding the most cost effective mechanisms to deliver it or of the added value of integrating treatment of acute malnutrition with treatment of common childhood illness and/or extensive communitybased nutritional program.

HYPOTHESIS:

Provision of SAM treatment at household level in a community through lady health workers will be as effective (recovery rate, survival, cost effectiveness, coverage) as treatment provided at facility level.

RESEARCH QUESTION:

Will SAM treatment delivered through LHW at household level be as effective as SAM treatment delivered at facility level by health center staff?

PRIMARY OBJECTIVES:

To evaluate the effectiveness (rate of recovery, relapse & coverage), of SAM treatment of children 6-59 months delivered at household level by first level health care providers (Lady health workers) compared with the standard CMAM program delivered at health facility by Government and ACF staff. To evaluate the cost effectiveness of treatment of SAM provided by LHWs at community level versus treatment delivered at health facility by Government and ACF staff.

SECONDARY OBJECTIVES:

To evaluate the characterization of the breast feeding and complementary feeding practices in both study arms. To identify the main socio-economic characteristics of the households in both study arms.

STUDY DESIGN:

The study will be a 2-armed cluster randomized controlled trial targeting children 60-59 months and their mothers for the treatment and prevention of acute severe malnutrition in children. Each cluster will be allocated to intervention group A, or control group B.

Cost-effectiveness analysis:

Cost effectiveness will be calculated to reflect the full range of resources required by service providers and households. A societal perspective will be taken with data collected on household costs incurred for participation in community and facility based activities. The approach will capture all resources used regardless of who incurs them, as used for cost analysis of other similar programs. Costs will be calculated with a combination of accounting records and estimates derived with an "ingredients" approach, using unit costs and quantities of inputs. Institutional costs will be estimated via accounting records. Costs which are known to be incurred by the program but which are not reflected in the accounting records (e.g. staff whose salaries are on different budgets, storage space which was not planned for in the original budget, etc.) will be estimated after identifying these costs through discussion with staff and document review. This data will be supplemented with costs calculated via an ingredients approach. Key informant interviews will be held with all key implementing staff to estimate their time allocation to project activities, in order to perform an activity based cost analysis.

Coverage assessment:

Coverage Assessments will be implemented in the two areas at the start the study, at six months of the study beginning and at the end of the study. SQUEAC methodology will be used. Coverage assessments are of particular interest in order to access the population that is not accessing treatment and understand its barriers to access. These assessments will be carried out by trained ACF staff.

MAIN STUDY OUTCOMES:

The key indicators to be captured are:

1. Effectiveness - recovery rate (proportion of cured children among SAM enrolled), supplement compliance rate, defaulter rate, relapse rate, Length of stay, average weight gain, hospital admission, and complications
2. Coverage rates and barriers to access (estimated using the SQUEAC methodology)
3. Health & Nutrition status of children (prevalence of malnutrition etc.)
4. Cost-effectiveness
5. Descriptive analysis to assess the distribution of various factors within and between groups, cluster-adjusted analyses will compare SAM rates (recovery, survival, relapse, default) observed in the different arms. Kaplan Meier statistics will be used for the comparison of post-treatment survival.

SAMPLE SIZE & RANDOMIZATION:

Investigators have calculated the sample size on the basis of SAM as the primary indicator; Investigators took 6% prevalence to calculate the sample size with an expected reduction of 20%. A sample size of 3 clusters per group with 150 individuals per cluster achieves 98% power to detect a difference of 0.200 between the group means when the standard deviation is 0.500 and the intracluster correlation is 0.00100 using a Two-Sided T-test with a significance level of 0.05000.

Definition of cluster:

A union council has been defined as the CLUSTER for the trial, a union council is the smallest administrative unit in the district which usually have a population of about 25000 to 30000, and this population has about 2500-3000 under five children, if Investigators consider the national rates of SAM in Pakistan which is about 6% Investigators will find more than 150 cases of SAM from each union council during the study period which will be enough sample to achieve the objectives of the trial. One union council has usually one health facility Basic health Unit (BHU) or Rural Health Center.

STUDY SITE:

The study will be carried out in Dadu district, a rural district of Sindh province of Pakistan. This district has been selected due to the high global acute malnutrition (GAM) rates, being affected by emergencies. Currently in Sindh, SAM treatment is delivered at health facility level.

BENEFICIARIES:

Main target beneficiaries would be children 6- 59 months of age fulfilling the case definition of severe malnutrition and their mothers.

DELIVERY OF INTERVENTION:

Intervention Arm (A): Lady Health Workers operating at field level in study arm A will be trained at the start of the study. The same training package will be delivered to all LHWs involved in the study regardless of their previous training and the trainings will be delivered by the Department of Health (once officially agreed), by ACF & AKU. All eligible children in the LHW´s catchment area will be identified and registered by the LHWs as part of their routine activities. In Pakistan national guidelines, SAM treatment admission criteria is MUAC <11.5 cm. Children 6- 59 months, with MUAC less than 11.5 cm and meeting eligibility criteria will be enrolled after obtaining consent and provide treatment of SAM at home and IYCF counseling and follow up till recovery. Children 60-59 months in the criteria for stabilization care will also be referred by the LHW.

The LHW will visit fortnightly to follow up all recruited children with SAM and receiving RUTF in their catchment population. If the child gets severely ill or having any complication the LHW will immediately refer that child to the nearest health facility for hospital based care. The LHW will record MUAC measurements on fortnightly follow up visits and weight and height will be recorded by the data collectors. Control Arm (B): Lady Health Workers operating at field level in study arm B will perform monthly home visit and will recruit and register all eligible children in their catchment area as part of their routine activities. The LHW will identify cases of SAM as per national CMAM guidelines through MUAC measurements and refer them to the nearest health facility where ACF staff will provide treatment in the facility as per standard CMAM guidelines.

DATA COLLECTION:

Data will be collected by an independent team, and not by LHWs. Data collection team will consist of 2 data collectors and a team leader. Data collectors and team leaders will be hired and trained to collect data by the study team.The team will visit identified households and the data will cross validate the LHW activities. The study team will collect information regarding children with SAM at baseline survey and during the study from LHWs and health facilities staff. A trained community health worker will visit the household having child with SAM and will take informed consent and recruit the child in the study.

Baseline Cross Sectional Survey :

A cross sectional survey will be conducted at household level in both arms

Fortnightly follow-up visits :

A fortnightly follow up of children will be carried out by the community health worker until the recovery of child this may takes up to 3-6 months during the first 3 months of the study , the purpose of this follow up is to collect the information regarding, acceptability, compliance, concurrent morbidities if any and record anthropometry (only weight & MUAC).

Monthly follow-up visits:

Monthly follow ups will be done by data collectors to capture the information on recovery, feeding practices, child's nutritional status morbidities & mortality. These follow ups will be continued for 6 months from the time of recruitment. Complete anthropometry (MUAC, Height and Weight) will be carried out during monthly follow ups.

Household cost survey:

Towards the end of the intervention, a household survey will be implemented on a random sample of program beneficiaries in both study areas to collect information on the direct and indirect costs they incurred in participating in the program. This will include information on cost of transportation, foods and medicines purchased, and time spent in accessing care.

ELIGIBILITY:
Inclusion Criteria:

* Born in the study area
* Presence of severe acute malnutrition (SAM).
* Ability of the parents or guardians to provide informed consent.

Exclusion Criteria:

* Presence of chronic debilitating illness.
* Residence outside of study areas.
* Inability or refusal of the parents or guardians to give informed consent, or refusal of assessment.
* Internally displaced population

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 762 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
To evaluate rate of recovery | 18 months
  To evaluate the rate of recovery of SAM treatment of children 6-59 months old delivered at household level by first level health care providers (Lady Health workers) compared with the standard CMAM program delivered at health facility by Govt and ACF staff.
  Pakistan national guidelines for the community based management of acute malnutrition 2014 will be used to measure this outcome.

SECONDARY OUTCOMES:
Prevalence of malnutrition | 18 months
  It will be estimated through cross sectional surveys.
To evaluate the cost effectiveness of treatment. | 18 months
  To evaluate the cost effectiveness of treatment of SAM provided by LHWs at community level versus treatment delivered at health facility by Govt and ACF staff.
Relapse from severe acute malnutrition | 18 months
  To evaluate the relapse of SAM treatment of children 6-59 months old delivered at household level by first level health care providers (Lady Health workers) compared with the standard CMAM program delivered at health facility by Govt and ACF staff.
  Pakistan national guidelines for the community based management of acute malnutrition 2014 will be used to measure this outcome.
Default cases of SAM | 18 months
  Pakistan national guidelines for the community based management of acute malnutrition 2014 will be used to measure this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sajid Soofi, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Project Office, Khairpur Nathan Shah, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bhutta ZA, Das JK, Rizvi A, Gaffey MF, Walker N, Horton S, Webb P, Lartey A, Black RE; Lancet Nutrition Interventions Review Group, the Maternal and Child Nutrition Study Group. Evidence-based interventions for improvement of maternal and child nutrition: what can be done and at what cost? Lancet. 2013 Aug 3;382(9890):452-477. doi: 10.1016/S0140-6736(13)60996-4. Epub 2013 Jun 6. PMID 23746776
- [Derived] Rogers E, Guerrero S, Kumar D, Soofi S, Fazal S, Martinez K, Moran JLA, Puett C. Evaluation of the cost-effectiveness of the treatment of uncomplicated severe acute malnutrition by lady health workers as compared to an outpatient therapeutic feeding programme in Sindh Province, Pakistan. BMC Public Health. 2019 Jan 17;19(1):84. doi: 10.1186/s12889-018-6382-9. PMID 30654780